CLINICAL TRIAL: NCT01028066
Title: Feeding Education in Patients Submitted to Percutaneous Transluminal Coronary Angioplasty: Randomized Clinical Trial
Brief Title: Feeding Education in Patients Submitted to Coronary Angioplasty
Acronym: PTCA-Nutri
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Moacyr Roberto Cucê Nobre, Heart Institute (InCor) HCFMUSP
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CAPPesq 0443/07; FAPESP 2007/54652-8
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2009-12

CONDITIONS: Coronary Angioplasty; Coronary Disease
Keywords: nutritional intervention; nutritional counseling; feeding behavior; food consumption; angioplasty
MeSH Terms: conditions — Coronary Disease; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional (Active Comparator): Traditional nutritional counseling
  Interventions: Other: Traditional
- Behavioral (Experimental): Dialogic nutritional counseling
  Interventions: Behavioral: Behavioral

INTERVENTIONS:
Other: Traditional — The control group will have access to the nutritionist to clear any doubts about the diet prescribed when went out the hospital and will be invited to attend a meeting nutrition in dialogic character at the end of 1 year to ensure fairness in action.
  Arms: Traditional
Behavioral: Behavioral — The intervention group will go through 4 meetings of food education, to be held within the institution, with approximately 1 hour long, composed of 3 to 8 patients, who may or may not be accompanied by a relative. The first three meetings will be monthly and the fourth will be 6 months after the last one. Each meeting will be developed within the context of dialogic and participatory education, directed to the adoption of a healthy diet and prevention and control of cardiovascular risk factors. The meetings will follow the order: Investigation, Contextualization, Awareness and Strengthening the nutritional concepts, according to the didactics of educator Paulo Freire.
  Arms: Behavioral

SUMMARY:
The simple knowledge that practices healthy lifestyle are important to reduce or prevent the progression of cardiovascular diseases it is not enough for effective changes accordingly. To nutritional education be successful, needs to promote changes in eating habits and not just transmit information. This is a behavioral intervention study in 200 consecutive patients submitted to percutaneous transluminary coronary angioplasty. The participants were randomized in two groups: intervention and control.

The intervention was a dialogic nutritional counseling and the control arm was a traditional nutritional counseling.

All participants will undergo long-term follow-up for cardiovascular events.

DETAILED DESCRIPTION:
Patients were hospitalized to realize elective coronary angioplasty in a especialized hospital in cardiovascular disease.

All data were obtained by a trained nutritionist.

ELIGIBILITY:
Inclusion Criteria:

* preserved cognitive status

Exclusion Criteria:

* no availability to attend the meetings of nutritional guidance

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-04; Primary Completion 2009-08 (Actual); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular event (new ptca, cabg, ischemic acute syndrome, myocardial infarction) and mortality (all causes) | 1 year (all outcomes) and 3 years (all outcomes)

SECONDARY OUTCOMES:
- Evaluate changes in eating habits, according to the transtheoretical model to adopt healthy eating habits - Check change in food intake - Identify the nutritional status and cardiovascular risk | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Moacyr Roberto Cucê Nobre, Principal Investigator — Heart Institute HCFMUSP
Locations (1):
- Heart Institute of Clinics Hospital of Medicine Faculty of São Paulo University, São Paulo, São Paulo, Brazil